CLINICAL TRIAL: NCT00886405
Title: Phase II Study That Evaluates Concurrent Chemotherapy and Radiotherapy With Nitroglycerin in Patients With Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Concurrent Chemotherapy and Radiotherapy With Nitroglycerin in Patients With Locally Advanced Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Oscar Arrieta Rodríguez, CONACYT
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB332/08; INCAN/CC/162/08; CA.030/CB332/08
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Locally Advanced Non Small-Cell Lung Canger
Keywords: Nitroglycerin; Locally advanced non small-cell lung cancer; Vascular endothelial growth factor; Hypoxia Inducible Factor; Clinical stage IIIA and/or IIIB (without pleural effusion)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nytroglicerin (Experimental)
  Interventions: Drug: Transdermal nitroglycerin

INTERVENTIONS:
Drug: Transdermal nitroglycerin — Transdermal nitroglycerin (25mg/day) during 5 days (2 days before and 3 days after chemotherapy) at the beginning of each chemotherapy cycle for a total of 4 cycles

SUMMARY:
Nitroglycerin will increase the effectiveness of treatment with induction chemotherapy and concurrent chemo-radiotherapy by reducing chemo-radio resistance through an increased oxygen pressure in tumoral tissue. The combination treatment of nitroglycerin and chemotherapy will result in longer disease-free and over-all survival in patients with locally advanced NSCLC

DETAILED DESCRIPTION:
Nitroglycerin decreases hypoxia-induced resistance to antitumor drugs due to inhibition of Hypoxia Inducible Factor alfa (HIF-1α), it increases oxygen pressure in tumoral tissue by augmenting tumor blood flow, increases apoptosis, activation of p53, and induces cellular growth inhibition. Randomized studies showed that the addition of transdermal nitroglycerin to non small cell lung cancer (NSCLC) patients with metastasis treated with vinorelbine and cisplatin achieved a significantly better global response to treatment than conventional treatment

ELIGIBILITY:
Inclusion Criteria:

* Histopathologic diagnosis of non small-cell lung cancer
* Clinical stage IIIA and/or IIIB without pleural effusion
* ECOG functional status 0 or 1
* No renal function alteration (GFR >50%)
* No hepatic function alteration (ALT and AST less than 2 times its normal value)
* Leucocytes more than 2,000/mcl
* Hemoglobin more than 10mg/dL
* Platelets more than 100,000/mcl

Exclusion Criteria:

* Ischemic heart disease
* Abnormal electrocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-04 (Actual); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Time to progression, over-all survival | 5 years

SECONDARY OUTCOMES:
Levels of oxidative stress through lipid peroxidation and quantification of VEGF Toxicity from treatment with chemotherapy and concurrent chemo-radiotherapy combined with transdermal nitroglycerin | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Oscar A Rodriguez, MD, Principal Investigator — National Counsil of Science and Technology
Locations (1):
- National Institute of Cancerología, Mexico City, Mexico City, Mexico